CLINICAL TRIAL: NCT03723720
Title: Calculating of Correlations Between ADR, PDR, MAP
Status: Completed | Type: Observational
Sponsor: Hospital Frydek-Mistek (Other)
Responsible Party: Principal Investigator, Ivana Mikoviny Kajzrlikova, MD, PhD, MD, Hospital Frydek-Mistek
Other Study IDs: MAP
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after colonoscopy over 50 years: All colonoscopies in patients over 50 years of age (screening, surveillance, diagnostic) excluding therapeutic, IBD, management of complications and sigmoidoscopies
  Interventions: Device: Colonoscopy

INTERVENTIONS:
Device: Colonoscopy — Endoscopic examination of large bowel

SUMMARY:
The aim of our study is to compare MAP (mean adenoma per colonoscopy) with ADR (adenoma detection rate) and PDR (polyp detection rate) of all colonoscopists in our department

DETAILED DESCRIPTION:
ADR (adenoma detection rate) is generally accepted quality indicator. For possible gaming with ADR other indicators are needed. MAP (mean adenoma per colonoscopy) reflects the quality of examination of entire colon and is considered to be the most objective quality indicator. The aim of our study is to compare MAP with ADR and PDR (polyp detection rate) of all colonoscopists in our department.

We want to retrospectively assess the quality indicators of all colonoscopies from January 2013 to December 2017. We want to calculate ADR, PDR and MAP of all our endoscopists for all colonoscopies in patients over 50 years of age excluding therapeutic, IBD, management of complications and sigmoidoscopies (screening, surveillance, diagnostic) and separately only for screening colonoscopies. Correlations between MAP/ADR and MAP/PDR will be performed using Pearson´s correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* people over 50 years of age coming for colonoscopic examination (screening, surveillance, diagnostic)

Exclusion Criteria:

* age under 50 years
* indication for colonoscopy: therapeutic, IBD, management of complications and sigmoidoscopies

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people over 50 years of age coming for colonoscopic examination
Sampling Method: Probability Sample
Enrollment: 6925 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
correlation between MAP and ADR for all and screening colonoscopies | january 2013 - december 2017
  Pearson´s correlation coefficient
correlation between MAP and PDR for all and screening colonoscopies | january 2013 - december 2017
  Pearson´s correlation coefficient
correlation between ADR and PDR for all and screening colonoscopies | january 2013 - december 2017
  Pearson´s correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Mikoviny Kajzrlikova, Principal Investigator — Doctor
Locations (1):
- Hospital Frydek-Mistek, Frýdek-Místek, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
ADR, PDR, MAP of all endoscopists in our unit for both all and screening colonoscopies